CLINICAL TRIAL: NCT05335954
Title: Phase 3 Therapeutic Interventional Study Evaluating the Efficacy of Noradrenaline in the Prevention of Hypotension Related to Intubation for Cardiac or Thoracic Surgery - Single-centre Prospective Randomised Controlled Study With Blinded Assessment of the Primary Endpoint
Brief Title: Therapeutic Study Evaluating the Efficacy of Noradrenaline in the Prevention of Hypotension Related to Intubation for Cardiac or Thoracic Surgery
Acronym: EPITUBE-HEART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC21_0144
Record Dates: First submitted 2021-11-09; First posted 2022-04-20 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Disorder; Hypotension
Keywords: general anesthesia; intubation; cardiac surgery; hypotension; noradrenaline
MeSH Terms: conditions — Heart Diseases; Hypotension | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient under anesthesia will not be aware of randomisation arm. the team collecting primary endpoint (hypotension under 55 mg during the 20 minutes after the start of anesthesia) will not be aware of patient assignation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noradrenaline (Experimental): Noradrenaline diluted to 16µg/ml infused at 0.06g/kg/min by peripheral venous line from the start of peripheral venous line from the start of preoxygenation
  Interventions: Drug: noradrenaline
- Standard care (No Intervention): standard care

INTERVENTIONS:
Drug: noradrenaline — noradrenaline
  Arms: Noradrenaline

SUMMARY:
Arterial hypotension during general anaesthesia (GA) is a serious event. While hypotension can occur during surgery, it usually occurs following induction of GA (i.e. following the injection of drugs to enable intubation). This is due to the injection of large doses of anaesthetic drugs with a vasodilatory effect over a short period of time to induce a deep sleep to allow intubation to take place for artificial ventilation.

The prevention of hypotension during surgery has been extensively studied. In contrast, the prevention of hypotension following GA induction has been the subject of only two randomised studies in the ICU and three non-randomised studies in the OR with small numbers of patients. The level of evidence for the use of noradrenaline in the operating theatre remains low.

The hypothesis of the study is that noradrenaline initiated during preoxygenation can reduce the incidence of hypotension during induction of general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Requiring cardiac or thoracic surgery under general anaesthesia
* Requiring a blood pressure catheter prior to GA induction

Exclusion Criteria:

* Hemodynamic instability on arrival in the operating room
* Hypotension on arrival in the operating theatre: Systolic blood pressure < 100 mmHg or Mean arterial pressure < 65 mmHg
* Hypertension on arrival at the operating theatre: Systolic blood pressure > 160 mmHg or Mean arterial pressure > 100 mmHg
* Adult under guardianship, curatorship or safeguard of justice
* Unable to give consent
* Pregnant or breastfeeding woman
* Emergency surgery (cannot be delayed by 24 hours)
* Current participation in an interventional protocol that interferes with the evaluation criteria of the study
* Not affiliated to or not benefiting from a social security scheme
* Lack of informed and written consent from the patient
* Patient with a dilated aorta with a risk of rupture (e.g. chronic dissection for example)
* Patient with severe aortic insufficiency
* Treated hypertensive history that may have hypersensitivity to noradrenaline and hypertensive flares hypertensive attacks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Intubation-related hypotension | Within 20 minutes of the start of general anesthesia (induction)
  Occurrence of at least one episode of arterial hypotension defined by a Mean Arterial Pressure below 55 mmHg with Mean Blood Pressure = (Systolic Blood pressure + 2xDiastolic Blood Pressure)/3

SECONDARY OUTCOMES:
Occurrence of complications | Within 20 minutes of the start of the intubation
  Occurrence (yes/no) of complications related to the intubation:
  Desaturation < 80%, Severe hypotension (defined as hypotension with systolic blood pressure < 80mmHg), Cardiac arrest, Death during intubation, Difficult intubation (more than two laryngoscopies and/or the use of an alternative technique after optimization of head position, with or without external laryngeal manipulation), Heart rhythm disorder (ventricular extrasystole, ventricular fibrillation, ventricular tachycardia) Esophageal intubation, Regurgitation/inhalation, Tooth breakage
Total dose of vasopressor | Within 20 minutes of the start of the intubation
  Total dose of vasopressors (noradrenaline, ephedrine, neosynephrine)
Duration of episodes of hypotension | Within 20 minutes of the start of the intubation
  Cumulative duration of episodes of hypotension < 55mmHg
Hypotension event | Within 20 minutes of the start of the intubation
  At least one Mean Arterial Pressure measurement < 65 mmHg
Hypertension event | Within 20 minutes of the start of the intubation
  At least one Systolic Blood Pressure measurement > 160 mmHg or Mean Arterial Pressure > 100mmHg
ECC Cardiac Output | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation generated Cardiac Output frequency in bpm (beat per minute)
ECC Arterial Line Pressure | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation generated Arterial Line Pressure in mmHg
ECC Arterial Line Temperature | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation generated Arterial Line Temperature in degree Celcius
ECC Mean Arterial Pressure | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation generated Mean Arterial Pressure in mmHg
ECC VO2 | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation generated VO2 (Volume O2) in Liter per Minute
ECC duration | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation duration in minutes
ECC SaO2 | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation generated SaO2 (Arterial Saturation in O2) in percentage
ECC SvO2 | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation generated SvO2 (Venous Saturation in O2) in percentage
ECC PaO2 | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation generated PaO2 (Arterial Pressure in O2) in kPa
ECC PaCO2 | Within 20 minutes of the start of the intubation
  Extra Corporeal Circulation generated PaCO2 (Arterial Pressure in CO2) in kPa
Delirium score | After extubation within 48 hours postoperatively
  At least episode with ICDSC (Intensive Care Delirium Screening Checklist) score of 4 or more (0 to 8, binary interpretation with scores from 0 to 4 excluding the presence of delirium and scores greater than or equal to 4 indicating the presence of delirium, the highest scores are not related with greater intensity of delirium)
Duration of Noradrenaline and Dobutamine treatments | Within 28 days after surgery
  Duration of treatment with Noradrenaline (in hours) and Dobutamine (in hours)
PaO2/FiO2 | In the 5 post-operative days
  Lowest value of PaO2/FiO2 (Arterial Pressure of O2 / Fraction inspired in Oxygen) measured
Dialysis | Within 28 days after surgery
  Use of dialysis in intensive care (Yes/No)
Hemolysis index | In the 5 post-operative days
  Maximum hemolysis index (0 to 10000, with higher scores being more pejorative)
Acute renal failure | In the 5 post-operative days
  Occurrence of acute renal failure. This criterion will be assessed using the KDIGO (Kidney Disease: Improving Global Outcomes) scale (stage 1 to 3 with higher stages being more pejorative). Any renal attack defined as at least stage I according to this classification (1.5 to 1.9 times the base rate) will be considered as acute renal failure. The "urinary output assessment" component of the KDIGO scale will not be used because of the frequency of use of diuretics in cardiac surgery.
CVA | In the 5 post-operative days
  Occurrence of a CVA (cerebrovascular accident)
Postoperative invasive ventilation duration | Until 28 days after surgery
  Duration of postoperative invasive ventilation in hours: this duration is defined by the duration of mechanical ventilation between arrival in intensive care and extubation
Stay in intensive care duration | Until 28 days after surgery
  Length of stay in intensive care in days: this duration is evaluated between the day of arrival in intensive care and the date on which the patient is considered to have left intensive care (no longer subject to monitoring in intensive care).
Hospitalization duration | Until 28 days after surgery
  Length of hospitalization in days
Mortality | Until 28 days after surgery
  Death of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Mickael VOURC'H, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Chu de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaillard C, Breul L, Foucher A, Rigal JC, David CH, Souab F, Canevet M, Ryan M, Bailly A, Morin H, Cadiet J, Geay C, Rozec B, Vourc'h M. Prophylactic norepinephrine infusion to reduce severe hypotension during induction of anaesthesia in patients undergoing cardiac surgery: a randomised controlled single-centre clinical trial. Br J Anaesth. 2025 Dec 10:S0007-0912(25)00795-0. doi: 10.1016/j.bja.2025.10.055. Online ahead of print. PMID 41381314